CLINICAL TRIAL: NCT00481715
Title: Interventions to Control Obesity in Colleges
Brief Title: Comparison of Two Workplace-Sponsored Obesity Prevention Programs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Laura Linnan, ScD/Associate Professor, UNC Chapel Hill
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 473; R01HL080656-01A1 (NIH)
Record Dates: First submitted 2007-05-31; First posted 2007-06-04 (Estimated); Last update posted 2011-01-27 (Estimated); Status verified 2011-01

CONDITIONS: Weight Loss
Keywords: Web-Based Weight Loss Program; Cash Incentive Weight Loss Program; North Carolina
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental): Web-based weight loss program
  Interventions: Behavioral: Web-Based Weight Loss Program
- 2 (Experimental): Cash incentive weight loss program
  Interventions: Behavioral: Cash Incentive Weight Loss Program
- 3 (Experimental): Web-based program plus the cash incentive program
  Interventions: Behavioral: Web-Based Weight Loss Program; Behavioral: Cash Incentive Weight Loss Program
- 4 (No Intervention): No intervention

INTERVENTIONS:
Behavioral: Web-Based Weight Loss Program — Participants will take part in a Web-based weight loss program.
  Arms: 1; 3
Behavioral: Cash Incentive Weight Loss Program — Participants will take part in a cash incentive weight loss program.
  Arms: 2; 3

SUMMARY:
Obesity has reached epidemic proportions in the United States with nearly 64% of American adults considered overweight or obese. Weight loss programs that take place at work have proven to be effective at promoting healthy lifestyles. The purpose of this study is to compare the effectiveness of a Web-based weight loss program versus a cash incentive weight loss program among employees at North Carolina universities and colleges.

DETAILED DESCRIPTION:
Obesity, which leads to higher rates of diabetes, cancer, and heart disease, is an increasingly important public health problem. Evidence suggests that the effects of poor diet and physical inactivity will soon overtake smoking as the leading cause of death. Obesity-attributable medical expenses account for 9.1% of the total annual medical expenditures in the United States, and may be as high as $78.5 billion. In North Carolina, obesity accounts for more than $2 billion annually in increased medical spending and nearly half of this total is financed through employer-provided health insurance. Weight loss programs that take place at work have demonstrated the ability to improve both employee health and the financial health of the company. However, few weight loss programs have been evaluated and implemented in the workplace. The purpose of this study is to compare the effectiveness of a Web-based weight loss program versus a cash incentive weight loss program among employees at universities and colleges in North Carolina.

This study will enroll approximately 1200 employees from 12 universities and colleges in North Carolina. Each university or college will be randomly assigned to one of the following four groups: 1) a Web-based weight loss program, 2) a cash incentive weight loss program, 3) the Web-based program plus the cash incentive program, or 4) neither program. Participants in the Web-based weight loss program will take part in a weekly Web-based weight control program that is comprehensive, individually focused, self-directed, and includes both weight loss and weight gain prevention information. In the cash incentive program, participants will receive a cash payment if they lose a pre-determined amount of weight at each follow-up weigh in. At baseline and Months 3, 6, 12, and 18, all participants will be weighed, body fat measurements will occur, and information on physical activity levels, eating behaviors, quality of life, work productivity, and medical expenses will be collected. During this study, study researchers will also monitor changes that occur in the physical and social environment on campus.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) greater than or equal to 25
* Current FT employee and member of the State Health Plan in North Carolina

Exclusion Criteria:

* Pregnant or breastfeeding
* Type 1 diabetes
* Currently taking weight loss medication
* Lacks internet access at work or home
* Previous weight loss surgery or plans to have weight loss surgery
* Answers "Yes" to any of the Physical Activity Readiness Questionnaire questions
* Known history of stroke, coronary heart disease, or type 2 diabetes, or possesses a BMI of 42 or higher AND does not have a medical clearance from a physician

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1020 (Actual)
Dates: Start 2008-09; Primary Completion 2010-05 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Weight loss | Measured at Mo 3,6, 12, 18 mo; powered at 12 mo measure

SECONDARY OUTCOMES:
Percentage of body fat; moderate physical activity (PA); moderate/vigorous PA and step counts; total calories consumed; fruits and vegetables consumed; total and saturated fat consumed; overall eating behavior; health related quality of life | Measured at Mo 3, 6, 12 and 18 mo
Self-reported health; presenteeism; productivity/work limits; turnover/absenteeism; medical expenditures data; campus changes in the physical/social environment | Measured at Mo 3, 6, 12, 18 mo

CONTACTS AND LOCATIONS:
Overall Officials: Laura A. Linnan, ScD, CHES, Principal Investigator — University of North Carolina, Chapel Hill